CLINICAL TRIAL: NCT05507177
Title: Effects of Communication Training to Involve Older People in Decisions to DEPRESCRIBE Cardiometabolic Medication: a Cluster-randomized Trial in Primary Care
Acronym: CO-DEPRESCRIBE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10506; 10140022010002 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Deprescriptions; Polypharmacy; Primary Health Care; Community Pharmacy Services; Decision Making, Shared
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Intervention Model Description: First healthcare provider teams are recruited. After inclusion, a team is randomly allocated the group I (intervention, receiving a training before conducting medication reviews) or group II (control group, receiving training after conducting medication reviews). After the teams in group I have been trained, teams in both arms will conduct ten medication reviews per team in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): patients that are treated in group I receive a medication review from healthcare providers that have already received the communication training programme
  Interventions: Other: communication training programme for healthcare providers
- Group II (No Intervention): patients that are treated in group II receive a medication review from healthcare providers that have not yet received the communication training programme

INTERVENTIONS:
Other: communication training programme for healthcare providers — the communication training programme is specifically designed to help Dutch primary care healthcare providers facilitate adequately deprescribing cardiometabolic medication in older patients
  Arms: Group I

SUMMARY:
The researchers will investigate the effects of a communication training for community pharmacists and general physicians that aims to make it easier for them to stop or lower medication for cardiovascular disease and/or diabetes in older patients.

The researchers expect that trained community pharmacists and general physicians will stop or lower medication for cardiovascular disease and/or diabetes in more patients compared to untrained community pharmacists and general physicians.

The researchers will recruit local teams consisting of a community pharmacist and one or more general physician, and allocate each team to either group I or group II. All teams in group I are first being trained, before they conduct a study-specific clinical medication review in 10 patients per team. All teams in group II will first conduct a more general clinical medication review in 10 patients per team too, before receiving the training. Patients will only be included after meeting in- and exlcusion criteria and signing an informed consent form. During the conduct of the study, the researchers will collect patient reported data and data on the conduct of the medication reviews. Retrospectively, the researchers will also collect data on the medication use of the patients from the pharmacy information system and specific medical data related to cardiometabolic disease of the patients from the physician's information system. The researchers will also assess the total costs and benefits of the intervention, and evaluate the training for the purpose of future implementation.

DETAILED DESCRIPTION:
RESEARCH QUESTION: The researchers will investigate the effects of a communication training program for community pharmacists and general physicians, that aims to facilitate stopping or lowering the prescription of medication for cardiovascular disease and/or diabetes in older patients.

HYPOTHESIS: The researchers expect that the training program will lead to more proactive stopping or lowering the prescription of medication for cardiovascular disease and/or diabetes, and that patients will be more involved in the decision to stop or lower.

STUDY DESIGN: The researchers will conduct a cluster-randomized trial in which 44 pharmacist-general practice teams in the Netherlands will be randomized to conducting medication reviews with 10 eligible patients as usual (control) or after receiving the deprescribing communication training program (intervention). STUDY POPULATION: People of 75 years and older using specific cardiometabolic medication and eligible for a medication review in The Netherlands will be included.

INTERVENTION: The training program is based on previous work and applies models for patient-centered communication and shared decision making. The training consists of 5 modules with supportive tools.

OUTCOME MEASURES: Primary outcome is the proportion of patients with deintensified cardiometabolic medication.

Secondary outcomes include patient involvement in decision-making, healthcare professional communication skills assessed by the patient, medication-related outcomes, attitudes towards deprescribing, medication regimen complexity and health-related quality of life. Additional safety and cost parameters will be collected.

SAMPLE SIZE/DATA-ANALYSIS: Based on a pilot study, the researchers have estimated that 167 patients are needed per study arm in the final intention-to-treat analysis using a mixed effects model. Taking loss to follow-up into account, 40 teams need to recruit 10 patients each. The researchers will conduct a baseline and a 6-months follow-up assessment, a process evaluation using the RE-AIM framework, and a cost effectiveness analysis.

ELIGIBILITY:
Inclusion criteria for the patients that receive a clinical medication review as part of the study:

* 75 years or older
* eligible for a clinical medication review according to the Dutch guidlines
* using one or more of the following medications:

  a) sulfonylurea derivative; (b) insulin; (c) any 2 glucose-regulating medications; (d) any 2 blood pressure-lowering medications; (e) statin
* managed and monitored by one of the participating HCP teams

Exclusion criteria for the patients that receive a clinical medication review as part of the study:

* diagnosed with type I diabetes
* not understanding Dutch language
* not giving or not able to give informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
proportion of patients in which one or more cardiometabolic medications is deprescribed | collected retrospectively, 6 months after the start of the medication review
  proportion of patients per study arm in which one or more medications for diabetes or cardiovascular disease has been lowered or stopped

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Stuijt PJC, Heringa M, van Dijk L, Faber A, Burgers JS, Feenstra TL, Taxis K, Denig P. Effects of a multicomponent communication training to involve older people in decisions to DEPRESCRIBE cardiometabolic medication in primary care (CO-DEPRESCRIBE): protocol for a cluster randomized controlled trial with embedded process and economic evaluation. BMC Prim Care. 2024 Jun 11;25(1):210. doi: 10.1186/s12875-024-02465-7. PMID 38862899